CLINICAL TRIAL: NCT02947672
Title: Effect of Intravenous Versus Intra-peritoneal Dexamethasone on the Incidence of Postoperative Nausea and Vomiting Following Laparoscopic Gynecological Surgeries
Brief Title: Intravenous Versus Intra-peritoneal Dexamethasone on the Incidence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01003060377
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Intravenous dexamethasone (Active Comparator): 50 patients will receive intravenous dexamethasone
  Interventions: Drug: Intravenous Dexamethasone
- Intra peritoneal dexamethasone (Active Comparator): 50 patients will receive intraperitoneal dexamethasone
  Interventions: Drug: Intraperitoneal Dexamesathone

INTERVENTIONS:
Drug: Intravenous Dexamethasone
  Arms: Intravenous dexamethasone
Drug: Intraperitoneal Dexamesathone
  Arms: Intra peritoneal dexamethasone

SUMMARY:
Effect of intravenous versus intra-peritoneal dexamethasone on the incidence of postoperative nausea and vomiting following Laparoscopic gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female patients
2. American society of anesthesiologist class I & II
3. Undergoing Laparoscopic gynecological surgeries

Exclusion Criteria:

1. Patient refusal to participate in the study
2. Patients with coagulopathy or under anticoagulation therapy.
3. Infection near the site of needle insertion.
4. Body mass index > 40kg/m2
5. Patients with any neurological or neuromuscular disorder or history of seizures.
6. Known allergy to any drug used in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 hours
  PONV will be measured by using Verbal Descriptive Scale

SECONDARY OUTCOMES:
Pain | 24 hours
  Pain will be assessed by using visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt